CLINICAL TRIAL: NCT06689202
Title: Assessment of Oral Health Knowledge, Attitude and Behavior of Adult Patients Attending a Dental School Hospital in Egypt: A Cross-sectional Study
Brief Title: Assessment of Oral Health Knowledge, Attitude and Behavior of Adult Patients in Egypt
Status: Completed | Type: Observational
Sponsor: NewGiza University (Other)
Responsible Party: Principal Investigator, Menna Nagy Sharkawy, Principle Investigator, NewGiza University
Other Study IDs: Knowledge,Attitude,Behavior
Record Dates: First submitted 2024-11-12; First posted 2024-11-14 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Oral Health Knowledge, Attitude and Practice Among Patients
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: The Hiroshima University - Dental Behavioral Inventory (HU-DBI) by Kawamura will be used as a validated instrument to assess oral health-related knowledge, attitudes, and behaviors (KAB). — The assessment will include 20 HU-DBI items, which employ a dichotomous response format (agree/disagree). However, only 12 items will be used to calculate the overall KAB score, which will range from 0 to 12, with higher scores indicating better oral health KAB.
Other: The Hiroshima University - Dental Behavioral Inventory (HU-DBI) by Kawamura will be used as a validated instrument to assess oral health-related knowledge, attitudes, and behaviors (KAB) — The assessment will include 20 HU-DBI items, which employ a dichotomous response format (agree/disagree). However, only 12 items will be used to calculate the overall KAB score, which will range from 0 to 12, with higher scores indicating better oral health KAB.

SUMMARY:
Oral health is a significant contributor to public health and is classified by the World Health Organization (WHO) as a major global health concern. Notably, one in two adults suffer from dental decay ,with oral diseases ranking among the most prevalent non-communicable disease (NCDs) . Thus, public health programs focus on modifying lifestyle factors for prevention rather than treatment. In developed countries , public health programs have successfully improved oral health through dietary and lifestyle modifications, as well as fluoride use .

Furthermore, oral health professionals have a crucial in role in influencing the behaviors of their patients and preventing oral diseases .Therefore, enhancing oral health knowledge is essential for positive health behaviors and hence better oral health outcomes .

ELIGIBILITY:
Inclusion criteria:

* Adult patients attending the diagnostic center in Newgiza University
* 18 years or older Exclusion criteria
* Patients who refuse to consent to participate in the survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients attending the diagnostic center in Newgiza University
Sampling Method: Non-Probability Sample
Enrollment: 288 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-03-25 (Actual); Study Completion 2025-05-10 (Actual)

PRIMARY OUTCOMES:
Oral Health Knowledge, Attitude & Behavior | November 2024-January 2025
  The overall KAB score is calculated using the 12 questions (Questions 2, 4, 6, 8, 9, 10, 11, 12, 14, 15, 16, and 19), with scoring as follows:
  * (A) indicates 1 point for the answer "Agree" to items (Questions 4, 9, 11, 12, 16, and 19).
  * (D) indicates 1 point for the answer "Disagree" to items (Questions 2, 6, 8, 10, 14, and 15).
  The KAB score ranges from 0 to 12, with higher scores indicating better oral health knowledge, attitudes, and behaviors. The scores are calculated as follows:
  1. The Knowledge (K) index score is derived from items 2, 8, 10, 15, and 19.
  2. The Attitude (A) index score is based on items 6, 11, and 14.
  3. The Behavior (B) index score is determined from items 4, 9, 12, and 16.

SECONDARY OUTCOMES:
DMFT Scores | November 2024-January 2025

CONTACTS AND LOCATIONS:
Locations (1):
- Newgiza University, Giza, Newgiza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sharkawy MN, Shaalan O. Oral health knowledge, attitudes, and behaviors of adult patients attending a dental school hospital in Egypt: a cross-sectional study. Sci Rep. 2025 Dec 5;15(1):43274. doi: 10.1038/s41598-025-29251-4. PMID 41350351